CLINICAL TRIAL: NCT06212869
Title: Green Light and Transcranial Direct Current Stimulation in Migraine Patients; a Randomized Control Trial.
Brief Title: Green Light and Transcranial Direct Current Stimulation in Migraine Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC01726 Amna Mehmood
Record Dates: First submitted 2023-12-19; First posted 2024-01-19 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Migraine
Keywords: migraine; green light; transcranial direct current stimulation
MeSH Terms: conditions — Migraine Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tDCS Group (Experimental): active tDCS with the prescribed medications for 20 minute. The intervention will conduct 3 consecutive days in a week.
  Interventions: Device: Transcranial direct current stimulation
- Sham tDCS Group (Sham Comparator): sham tDCS with the prescribed medications for 20 minute. The intervention will conduct 3 consecutive days in a week.
  Interventions: Device: Sham transcranial direct current stimulation
- Green Light Group (Experimental): green light exposure with the prescribed medications for 1-2 hour. The intervention will conduct 5 days in a week.
  Interventions: Device: Green light

INTERVENTIONS:
Device: Transcranial direct current stimulation — tDCS group will give active tDCS with the prescribed medications for 20 minute. The intervention will conduct 3 consecutive days in a week.
  Arms: tDCS Group
Device: Sham transcranial direct current stimulation — Sham tDCS group will give sham tDCS with the prescribed medications for 20 minute. The intervention will conduct 3 consecutive days in a week.
  Arms: Sham tDCS Group
Device: Green light — Green light group will give green light exposure with the prescribed medications for 1-2 hour. The intervention will conduct 5 days in a week.
  Arms: Green Light Group

SUMMARY:
There is a lack of evidence on the clinical outcome of green light exposure, as it is the emerging, novel proposal of treatment. There are a lot of researches present with small sample size which should be done on large population. In last conducted studies, session numbers of the applied modality are less. There is no comparison of tDCS with green light for migraine. The literature suggested the neuromodulation influenced by these interventions that may result in reduction of migraine.

DETAILED DESCRIPTION:
Migraine treatments encompass both medicinal options, such as acute and preventive medications, as well as a variety of non-pharmacological therapies. The range of acute medications that are available can be categorized into four different treatment approaches for treating mild to moderate-severity attacks, which involve the use of acetaminophen and/or NSAIDs. For patients experiencing severe attacks or those who do not respond to the initial strategy, a triptan-based strategy is recommended. According to the American Academy of Neurology (AAN), there is strong supporting evidence for the effectiveness of several medications in preventing migraines, including metoprolol, timolol, propranolol, divalproex sodium, sodium valproate, and topiramate. There are some non-pharmacological approaches present like non-invasive and invasive neuromodulation. In non-invasive treatment, transcutaneous cranial nerve stimulation, vagus nerve stimulation, single-pulse transcranial magnetic stimulation (sTMS), transcranial direct current stimulation (tDCS), percutaneous mastoid stimulation and non-painful brachial electric stimulation are involved. In invasive neuromodulation, occipital nerve stimulation, sphenopalatine ganglion stimulation, and high cervical spine cord stimulation are involved.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria established by the International Headache Society,
* patient must have had at least 5 headache attacks that lasted 4-72 hours (untreated or unsuccessfully treated)
* headache must have had at least 2 of the following characteristic; Unilateral location & Pulsating quality,
* An average headache pain intensity of migraine episodes of ≥5 at numeric pain scale (NPS) over the 10 weeks prior to enrolling in the study.

Exclusion Criteria:

* Mental illness,
* Photophobic individual,
* Presence of shunt and/or implant at the cranial region,
* Brain tumors,
* Wound at skull

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Structured Headache Diary Data for frequency of migraine | Week 4
  diaries make it possible to record prospectively the characteristics of every attack and the use of headache calendars is indicated for evaluating the time pattern of headache, identifying aggravating factors and evaluating the efficacy of preventive treatment. This may reduce the recall bias and increase accuracy in the description.
Numeric Pain Scale (NPS) for intensity of migraine | Week 4
  NPS was implemented in clinical practice due to its rapidity both verbally and in writing. Due to its convenience, it is common for hospitals to measure pain using the 0 to 10 NPS scale.
Multidimensional pain inventory (MPI) for migraine impact | Week 4
  Multidimensional Pain Inventory (MPI) is one of the most widely used multidimensional instruments to measure adaptation to pain. It is a self-administered questionnaire comprising 12 empirically derived scales that measure dimensions of pain perception, life interference due to pain, perception of life control, affective distress, and social support. The instrument uses a clustering approach to derive three distinct subgroups: Dysfunctional (Dys), interpersonally distressed (ID), and adaptive copers (AC).

SECONDARY OUTCOMES:
Migraine-specific Quality of Life Survey (MSQ 2.1) for quality of life | Week 4
  The MSQOL is a measure to assess the effects of migraine over the longer term on patient well-being over a nonspecified time period, and the MQoLQ is designed to measure the short-term impact of migraine over a 24-hour period following the start of therapy for migraine.

CONTACTS AND LOCATIONS:
Overall Officials: Mirza Obaid Baig, MSPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferrari MD, Goadsby PJ, Burstein R, Kurth T, Ayata C, Charles A, Ashina M, van den Maagdenberg AMJM, Dodick DW. Migraine. Nat Rev Dis Primers. 2022 Jan 13;8(1):2. doi: 10.1038/s41572-021-00328-4. PMID 35027572
- [Background] Andreou AP, Edvinsson L. Mechanisms of migraine as a chronic evolutive condition. J Headache Pain. 2019 Dec 23;20(1):117. doi: 10.1186/s10194-019-1066-0. PMID 31870279
- [Background] Martin LF, Patwardhan AM, Jain SV, Salloum MM, Freeman J, Khanna R, Gannala P, Goel V, Jones-MacFarland FN, Killgore WD, Porreca F, Ibrahim MM. Evaluation of green light exposure on headache frequency and quality of life in migraine patients: A preliminary one-way cross-over clinical trial. Cephalalgia. 2021 Feb;41(2):135-147. doi: 10.1177/0333102420956711. Epub 2020 Sep 9. PMID 32903062
- [Background] Puledda F, Silva EM, Suwanlaong K, Goadsby PJ. Migraine: from pathophysiology to treatment. J Neurol. 2023 Jul;270(7):3654-3666. doi: 10.1007/s00415-023-11706-1. Epub 2023 Apr 8. PMID 37029836
- [Background] Hussain G, Rasul A, Anwar H, Sohail MU, Kamran SKS, Baig SM, et al. Epidemiological data of neurological disorders in Pakistan and neighboring countries: a review. Pakistan Journal of Neurological Sciences (PJNS). 2017;12(4):52-70.